CLINICAL TRIAL: NCT04068350
Title: Epidemiological Study of Post-operative Chronic Pediatric Pain.
Acronym: PEDIACHRO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2009/18
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Pain; Postoperative Pain
Keywords: Pediatrics
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: The evaluation at 3 months of the postoperative pain will be carried out without the information collected in preoperative and immediate postoperative.
  Interventions: Other: Pain questionnaire

INTERVENTIONS:
Other: Pain questionnaire — Pain questionnaire, 3 months after surgery

SUMMARY:
This study aims to estimate prevalence and determine risk factors for chronic pain at 3 months post-operative in pediatric surgery.

DETAILED DESCRIPTION:
Chronic pain, defined as continuous or intermittent pain for 3 months or more, postoperative because in the territory of the surgical procedure and does not exist before the operation, is common in adults. Its prevalence varies according to the surgeries between 10 and 50% of the operated adults. The factors potentially responsible for their occurrence are gradually being highlighted in the recent literature, which has made it possible to develop an appropriate analgesic management strategy.

In pediatric surgery, acute pain has long been known and treated as early as possible using multimodal analgesic techniques. On the other hand, there are very few studies evaluating postoperative chronic pain 3 months after infant surgery, as was the case a few years ago in adults.

This study aims to estimate prevalence and determine risk factors for chronic pain at 3 months post-operative in pediatric surgery.

ELIGIBILITY:
Inclusion Criteria:

All children between the ages of 6 and 18, who are scheduled for surgery or video-surgery, scheduled or urgent, in the pediatric surgery department of the Bordeaux University Hospital.

All patients who consented to participate in the research.

Exclusion Criteria:

* All children operated on outpatient surgery.
* Children and parents with difficulties in understanding the questionnaires.
* Refusal of the child or one of the parents.
* Change of home planned during the post-operative follow-up period (3 months).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children between the ages of 6 and 18, who are scheduled for surgery or video-surgery, scheduled or urgent, in the pediatric surgery department of the Bordeaux University Hospital. The main interventions concerned by this protocol are:
  * Thoracotomies and thoracoscopies
  * Cholécysctectomie
  * Laparotomy and appendectomy
  * Inguinal surgery (inguinal hernia and testicular ectopia)
  * Orthopedic surgery
  * Urologic surgery (hypospadias, circumcision and upper urinary tract surgery)
Sampling Method: Non-Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2010-03-21 (Actual); Primary Completion 2011-12-21 (Actual); Study Completion 2011-12-21 (Actual)

PRIMARY OUTCOMES:
Chronic postoperative pain | 3 months after surgery
  Visual analogic scale from 0 to 100: (between 0 and 30: low pain, between 30 and 60: moderate pain, between 60 and 100: severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BATOZ, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No